CLINICAL TRIAL: NCT04155996
Title: Data Acquisition Study in Patients With Type 2 Diabetes Mellitus Who Are Inadequately Balanced With Oral Antidiabetic Agents and Basal Insulin
Brief Title: Data Acquisition Study in Inadequately Balanced Patients With Type 2 Diabetes Mellitus
Status: Terminated | Type: Observational
Why Stopped: Study terminated prematurely due to COVID-19 pandemic
Sponsor: ValoTec (Industry)
Collaborators: APHP (Other)
Responsible Party: Sponsor
Other Study IDs: VTC-MLS-EC01
Record Dates: First submitted 2018-06-22; First posted 2019-11-07 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- data collection: 20 patients
  Interventions: Device: data collection

INTERVENTIONS:
Device: data collection — Patients will receive a full data acquisition set with CGM sensors, an activity tracker and a smartphone application in which they can log daily events.

SUMMARY:
The aim of this study is to collect continuous glucose monitoring (CGM) data, coupled with physical activity and everyday day life data. The purpose of this data collection is to help diabetologists to make recommendations to optimize type 2 diabetic patient management.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patient (T2D) with HbA1c ≥ 8% in the month prior to inclusion
* Patient is treated with oral anti-diabetics and / or analogous combined with basal insulin therapy (1 injection of slow-acting insulin in the evening)
* Age ≥ 35 years
* Diabetes diagnosis done over 1 year ago
* Patient accepting for 2 periods of 14 days spaced at most 3 days to wear a Freestyle glucose meter, a bracelet for measuring physical activity and to log daily life events in a dedicated smartphone application
* Patient is able to use a smartphone
* Patient is affiliated to the French health insurance system

Exclusion Criteria:

* Patient has Type 1 diabetes, diabetes secondary to pancreatic pathology, endocrinopathy or iatrogenic diabetes
* Patient is treated with a rapid-acting insulin
* Patient has had a severe hypoglycaemia in the year preceding inclusion
* Patent has a severe renal insufficiency (defined by a Glomerular Filtration Rate below 30 ml/min)
* Patient has had a myocardial infarction or other life-threatening medical condition in the last 6 months
* Patient has cognitive disorders or evolutionary psychiatric pathology
* Pregnant woman or woman likely to be pregnant, breastfeeding woman
* Patient plans to travel outside europe during the study
* Patient is participating to another clinical study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetic patients followed by french primary care or specialized centers.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Data collection - Blood glucose levels | 28 days
  Patients wear a continuous glucose monitoring patch and record blood glucose level measurements (in mg/dl) over time.
Data collection - Number of steps | 28 days
  Patients wear an activity tracker that will record their number of steps over time.
Data collection - Sleep hours | 28 days
  Patients wear an activity tracker that will record their sleep hours (sleep start time and sleep end time) during nighttime.

SECONDARY OUTCOMES:
Data collection - Daily meals information | 28 days
  Patients manually record information about meals in a dedicated smartphone application.
  Each meal size (Small, Medium or Large) and glycemic index (Low, Medium or High) is evaluated by patients in the application.
Data collection - Physical activity information | 28 days
  Patients manually record information about physical activities in a dedicated smartphone application.
  Each physical activity duration (Short, Medium or Long) and intensity (Low, Medium or High) is evaluated by patients in the application.
Data collection - Medical treatment information | 28 days
  Patients manually record information their medical treatment in a dedicated smartphone application.
  Treatment intake times are recorded in the smartphone application.

CONTACTS AND LOCATIONS:
Overall Officials: Marine HALBRON, MD, Principal Investigator — APHP
Locations (1):
- GH Pitié Salpêtrière Charles Foix, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No